CLINICAL TRIAL: NCT03781921
Title: Disentangling Emotional Processing From Regulation in Bulimia Nervosa
Brief Title: The Neural Bases of Emotion Regulation in Bulimia Nervosa
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 1819/IRASLR-V/1
Record Dates: First submitted 2018-12-10; First posted 2018-12-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Bulimia Nervosa; Emotions; Emotional Impulsivity
Keywords: eating disorder; Electroencephalography; emotion regulation; emotion processing; negative urgency
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders; Emotional Regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BN: Females with a current diagnosis of Bulimia Nervosa between 18 and 50 years old
  Interventions: Other: No intervention
- Controls: Females with no current or past diagnosis of any eating disorder; between 18 and 50 years old
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention. Each group will conduct the same tasks and questionnaires and we will compare performances between groups.

SUMMARY:
This project aims to explore emotional processing and regulation in individuals with Bulimia Nervosa (BN) with a view to better understand its underlying causes. Previous research suggests that binge eating and purging behaviours may be linked to difficulties with emotions and impulses. However, most of the research has been conducted using self-report methods, despite the fact that these individuals have difficulties identifying and describing their emotions (known as alexithymia), making the use of self-report questionable. This project is the first to use electroencephalography (EEG) as an objective method to disentangle emotional processing and regulation in these individuals. A combination of three tasks and questionnaires will be used to measure various aspects of an emotional response and its link to impulsive behaviours in individuals with BN (N=35) and healthy controls (N=35). This study has the potential to inform future treatment for these individuals.

DETAILED DESCRIPTION:
Relevance:

Over 1.6 million people in the UK are affected by an eating disorder and approximately 40% of these - 640,000 - suffer from bulimia nervosa (BN). Research shows that at 10 years after diagnosis, only about half the people with BN will have recovered fully, demonstrating the importance of developing new and more effective treatment. A recently published study suggests that training emotion regulation skills may work as an alternative treatment. This is because difficulties with emotions have been shown to contribute to eating disorder pathologies. However, most studies looking at emotional difficulties in this population have used self-report methods, despite the fact that high levels of alexithymia (difficulties with identifying and describing emotions) characterise this population, indicating that these findings are potentially flawed. In addition, self-report data show that two processes seem involved in eating disorders, namely emotional intensity and emotional dysregulation. However, experiencing emotions with higher intensity also makes it harder to reappraise emotions so it is not clear whether individuals with BN actually have a real deficit in emotion regulation, because self-reports cannot distinguish the two. The current project is proposing to use an objective way to disentangle these aspects of emotional processing by looking at two brain activities. The first is called the N1 because it appears about 100 ms after the presentation of a stimulus and is of negative amplitude; the second is called the LPP for Late Positive Potential.

This proposal also aims to investigate the mechanisms behind the observed link between negative urgency (acting impulsively under distress) and binge eating by exploring the brain's ability to filter out irrelevant stimuli in the environment -also called sensory gating. Whilst individuals are constantly being stimulated by information, the brain usually filters irrelevant information to prevent the cortex from being overloaded. However, if too much attention is directed towards a stimulus (such as a negative event or food stimuli), sensory gating deficits may occur, which could lead to cognitive deficits such as negative urgency. In a previous study, the investigators have shown impaired sensory gating in bipolar disorders and due to similarities in affective processing between bipolar disorder and BN as well as high comorbidity between these disorders, the investigators suggest similar mechanisms may be in place in BN.

This project has strong implications for treatment, because different approaches could be used depending on what processes are affected (e.g. training to reallocate attention vs helping with emotion regulation strategies).

Research Questions:

This research aims to answer the following four research questions using three tasks to measure emotional processing and regulation (Task 1), emotional sensory gating (Task 2), and negative urgency (Task 3).

1. Is binge eating associated with higher emotional intensity, as indicated by larger N1 amplitudes in BN compared to controls?
2. Do individuals with BN show poor emotion regulation skills, as indicated by larger LPP amplitudes in the reappraisal condition compared to controls?
3. Do individuals with BN show impaired emotional sensory gating, as indicated by lower P50 ratio compared to controls? 3.1. If so, can deficits in emotional sensory gating explain the emotional difficulties seen in BN, including negative urgency?
4. To what extent do emotional intensity, emotion regulation deficits and emotional sensory gating deficits predict binge eating in BN?

Participant selection Since there are no similar studies conducted in participants with Bulimia Nervosa, the investigators calculated our sample size based on power analysis from other studies. Sample size varied between 13 and 33 participants to have an 80% chance of finding an effect and a level of significance of 5%. The investigators will recruit 35 participants in each group. Thirty five control participants will be recruited through a mailing list available at Bournemouth University (which includes students as well as non-students).

Thirty five female participants with bulimia nervosa (BN) will be recruited from Kimmeridge Court in Bournemouth. Dr Ciaran Newell (Consultant Nurse Eating Disorders) will advertise our study to new patients diagnosed with BN. When patients are referred to Kimmeridge court, they will be told about the current study. It will be emphasised that taking part in the study is completely separate from their treatment and that whether or not they decide to participate will not have any influence on their treatment. If participants decide to participate they will be told to contact the PI (Dr Laura Vuillier) who will give them more information over the phone or face to face, depending on their preferences.

Study Design If participants do agree to participate, participants will be sent a survey via email. At the start of the study, participants will see a participant information sheet detailing the study. Participants will then be asked to sign an electronic consent form if they agree to participate. This survey will ask questions about their emotions and their eating patterns. This survey will take approximately 30 minutes to complete. Their response will be pseudonymous as participants will be asked to enter a pseudonymous code. At the end of the survey participants will be asked to contact the experimenter to arrange a convenient time for the laboratory session.

The laboratory session will take about 3 hours, including breaks and will take place in the premises of Bournemouth University (Talbot campus). Thereparticipants will be given another information sheet detailing this next part of the study. Participants will be asked to sign another consent form before they can proceed. If participants agree to participate, the researcher will administrate a structural interview (using the SCID short version) to confirm their eating disorder diagnosis. After this, the electroencephalography (EEG) experiment will start. All parts of the experiment (including the survey, the SCID and the three tasks) will be pseudonymous and participants will not have to give any personal detail such as their name. The only place the investigators will ask for their name is when participants sign the consent form. However, these will be stored in a separate location and it will not be possible to link these with their data.

For the purposes of the experiment, a cap with electrodes will be placed on their head to record their brain activity. This will take about 30 minutes to set up. Then, participants will be asked to complete 3 computer tasks: an emotion regulation task (task 1), a sensory gating task (task 2) and a GoNogo task (task 3, all three are defined below). Each task will take approximately 30 minutes to complete. Participants will be told they can take a break during each task and also between tasks. Then the investigators will remove the cap with the electrodes and the participants will be able to wash their hair (some gel is used on the electrodes) before they leave.

Task 1: Emotional processing and regulation This task will show 50 emotional pictures from a picture library accompanied by a neutral or negative description. For instance, a picture of a woman dying will be either preceded by a neutral description (These doctors will save the woman's life) or negative description (These workers have found a war victim). Reappraisal is measured with the neutral description as participants will interpret the picture in a less negative way. Previous work conducted in healthy participants show a reduction in one brain activity (the LPP, or Late Positive Potential) in the reappraisal condition, and larger amplitudes for another brain activity (the N1, for Negative activity appearing 100ms after a stimulus) for stimuli with a negative valence reflecting higher attentional processes.

Task 2: Sensory gating The sensory gating deficit hypothesis will be tested in a paired-click paradigm using 40 pictures of negative valence, 40 pictures of food, and 40 neutral pictures from an affective picture library. Participants will be asked to passively watch the 120 pictures while the participants hear two clicks. Sensory gating will be measured as the difference in amplitude in one brain activity (called the P50) between the first and second click in all three conditions. This difference in amplitude shows that the brain filtered the second stimuli.

Task 3: Negative urgency Negative urgency will be measured with our GoNogo task. This task requires participants to 'go' (e.g. key press) when viewing a specific stimulus, but to 'not go' (e.g. not key press) when viewing a different stimulus. To provide the emotional context to our paradigm the task will use 50 negative emotional and 50 neutral pictorial stimuli. The percentage of false alarms is considered an index of negative urgency, since it represents an unsuccessful attempt at controlling an impulsive action.

Questionnaires:

The investigators will use validated questionnaires including the Eating Disorder Examination Questionnaire, the Difficulties in Emotion Regulation Scale, the Toronto Alexithymia Scale, and the Barratt Impulsiveness Scale to correlate self-report data with brain activity and understand how these levels of explanation are related.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Fluent in English
* With a diagnosis of bulimia nervosa for the BN group and without a diagnosis of any eating disorder for the control group

Exclusion Criteria:

* Males
* Under 18 or over 50

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only individuals being genetically females (As opposed to simply identifying as one) will be taking part in the study.
Study Population: Participants will be identified as they come to be diagnosed at Kimmeridge Court in Bournemouth, the local NHS clinic for people with eating disorders. Leaflets will be left in the waiting room area and their clinician will also give individual leaflets to individuals those patients meeting our inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
LPP | Only once on the day of the electroencephalography task
  Late Positive Potential differences in amplitude between the different groups and different conditions
N1 | Only once on the day of the electroencephalography task
  Differences in amplitude between the different groups and different conditions
P50 | Only once on the day of the electroencephalography task
  Differences in amplitude between the different groups and different conditions
False alarm rate | Only once on the day of the task
  Differences in rate between the different groups and different conditions

CONTACTS AND LOCATIONS:
Overall Officials: Laura Renshaw-Vuillier, PhD, Principal Investigator — Bournemouth University
Locations (2):
- United Kingdom (2):
  - Bournemouth University, Bournemouth
  - Dorset Healthcare University NHS Foundation Trust, Bournemouth

IPD SHARING:
Plan to Share IPD: Yes
Other researchers in the team will have access to the participant anonymised data for further analysis. This will be shared through a secure server.
  The anonymised data will also be saved on Bournemouth secured data repository for other researchers outside the research team to have access to it (requirement for publications etc)
Time Frame: The participant's anonymous data will be saved for 10 years on Bournemouth secured online data repository
Access Criteria: Anyone with the link will be able to acess the data. The link will be distributed during the publication process.